CLINICAL TRIAL: NCT07361679
Title: Combined Administration of Low Molecular Weight Heparin and Aspirin Versus Aspirin Alone in Gravidas at High Risk for Preeclampsia: A Randomized Controlled Trial
Brief Title: LDA and LMWH vs LDA Alone in High-risk Patients for Preeclampsia Prevention
Acronym: preGO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandra Hospital, Athens, Greece (Other)
Responsible Party: Principal Investigator, Georgios Daskalakis, Professor of Obstetrics and Gynecology, Alexandra Hospital, Athens, Greece
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 724/23-11-2022
Record Dates: First submitted 2025-12-21; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Preeclampsia Severe; Toxemia Of Pregnancy; Preeclampsia; Pregnancy Complications; Hypertension, Pregnancy-Induced; Gestational Hypertension
Keywords: preeclampsia; gestational hypertension; toxemia; Preeclampsia prevention; Low molecular weight heparin; tinzaparin; High-risk pregnancy; LMWH; Maternal-fetal medicine
MeSH Terms: conditions — Pre-Eclampsia; Pregnancy Complications; Hypertension, Pregnancy-Induced; Toxemia | interventions — Aspirin; Tinzaparin; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Intervention Model Description: Two parallel groups: Arm 1 receives aspirin alone, Arm 2 receives aspirin plus weight-adjusted LMWH
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin Alone (Active Comparator): Participants receive aspirin 160 mg orally once daily before bedtime from enrollment (<16 weeks gestation) until 36 weeks gestation.
  Interventions: Drug: Aspirin
- Aspirin plus LMWH (Experimental): Participants receive aspirin 160 mg orally once daily before bedtime PLUS weight-adjusted tinzaparin subcutaneously once daily in the morning (4,500 Anti-Xa IU for weight ≤60 kg, 6,000 Anti-Xa IU for weight 60-90 kg, 8,000 Anti-Xa IU for weight >90 kg) from enrollment (<16 weeks gestation) until 36 weeks gestation.
  Interventions: Drug: Aspirin; Drug: Tinzaparin

INTERVENTIONS:
Drug: Aspirin — Aspirin 160 mg orally once daily before bedtime. Duration: From enrollment (<16 weeks gestation) until 36 weeks gestation.
  Other Names: ASA; Low-dose aspirin; Acetylsalicylic acid
Drug: Tinzaparin — Weight-adjusted tinzaparin administered subcutaneously once daily in the morning: 4,500 Anti-Xa IU/day for weight ≤60 kg, 6,000 Anti-Xa IU/day for weight 60-90 kg, and 8,000 Anti-Xa IU/day for weight >90 kg. Duration: From enrollment (<16 weeks gestation) until 36 weeks gestation.
  Other Names: Low molecular weight heparin; Innohep; LMWH
  Arms: Aspirin plus LMWH

SUMMARY:
Preeclampsia is a major cause of maternal and perinatal morbidity and mortality worldwide. Low-dose aspirin started in the first trimester reduces the risk of preeclampsia in high-risk women. Low molecular weight heparin (LMWH) has shown potential benefits in addition to aspirin for preventing preeclampsia through its anticoagulant, anti-inflammatory, and endothelial protective effects. However, current evidence is limited and conflicting regarding the added value of LMWH to aspirin. This randomized controlled trial aims to evaluate the efficacy of combined aspirin and LMWH, compared to aspirin alone, for reducing the incidence of preeclampsia in high-risk gravidas.

DETAILED DESCRIPTION:
This is a prospective, randomized, single-center, open-label trial conducted at the First Obstetrics and Gynecology Clinic of Alexandra Hospital, Athens, Greece. One hundred pregnant women at high risk of preeclampsia (risk >1:150) will be randomly allocated 1:1 to receive either 160mg aspirin daily (n=50) or 160mg aspirin plus weight-adjusted therapeutic doses of LMWH (tinzaparin 4,500-8,000 IU daily based on weight) (n=50) initiated before 16 weeks gestation until 36 weeks.

Risk assessment will be performed using the internationally recognized FMF (Fetal Medicine Foundation) model, combining first trimester ultrasound examination, biochemical markers, and individual medical history.

The primary outcome is the incidence of preeclampsia. Secondary outcomes include development of early preeclampsia (<34 weeks), gestational hypertension, HELLP syndrome, spontaneous preterm labor, intrauterine growth restriction, placental abruption, and various neonatal outcomes.

Blood samples will be collected at 20-24, 32-34, and 36 weeks to measure biomarkers including PlGF, sFlt-1, E-Selectin, IL-1β, IL-6, IL-10, TNF-α, sFlt-1/PlGF ratio, and systemic immune-inflammation index (SII). Regular telephone follow-up will be conducted to monitor adherence and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* High risk for preeclampsia (risk >1:150) based on FMF screening algorithm combining first-trimester ultrasound, biochemical markers, and medical history
* Gestational age <16 weeks at enrollment
* Maternal age ≥18 years
* Willing and able to provide written informed consent
* Adequate ability for follow-up (direct telephone communication, accessible residence)

Exclusion Criteria:

* Multiple pregnancy
* Current permanent aspirin use for other medical indications
* Serious congenital fetal abnormality detected on ultrasound
* Contraindication to aspirin or low molecular weight heparin including: known hypersensitivity, active peptic ulcer disease, bleeding disorders or coagulopathy, severe thrombocytopenia (platelet count <100,000/μL), active or recent significant bleeding, history of heparin-induced thrombocytopenia
* Pre-existing severe renal failure (creatinine clearance <30 mL/min)
* Unable to provide informed consent
* Low probability of adequate follow-up (residence in remote areas without telephone access, accommodation in temporary structures)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Preeclampsia | From enrollment until delivery (up to 40 weeks gestation)
  Preeclampsia defined as gestational hypertension (BP ≥140/90 mmHg on at least two measurements ≥4 hours apart) after 20 weeks' gestation accompanied by one or more of: (1) Proteinuria (≥30 mg/mmol protein:creatinine ratio, ≥8 mg/mmol albumin:creatinine ratio, ≥0.3 g/24h, or ≥2+ dipstick); (2) Maternal end-organ dysfunction including neurological complications (severe headaches, visual scotomata, eclampsia, stroke, clonus), pulmonary oedema, haematological complications (platelet count <150,000/μL, disseminated intravascular coagulation, haemolysis), acute kidney injury (creatinine ≥90 μmol/L or 1 mg/dL), or liver involvement (elevated ALT or AST >40 IU/L); or (3) Uteroplacental dysfunction (fetal growth restriction, abnormal umbilical artery Doppler waveform analysis, placental abruption, angiogenic imbalance, or intrauterine fetal death), per ISSHP 2021 classification.

SECONDARY OUTCOMES:
Systemic Immune-Inflammation Index (SII) | At 20-24 weeks, 32-34 weeks, and 36 weeks gestation
  Systemic immune-inflammation index calculated as SII = P × N/L, where P, N, and L are the peripheral blood platelet count, neutrophil count, and lymphocyte count respectively (cells per liter)
Incidence of Preterm Preeclampsia | From enrollment until 37 weeks gestation
  Development of preeclampsia before 37 weeks gestation
Prevalence of placental histopathological lesions | At delivery
  Histopathological examination of placental tissue including assessment of maternal vascular malperfusion, fetal vascular malperfusion, villous lesions, inflammatory lesions, and other pathological findings according to standardized criteria
Soluble fms-like Tyrosine Kinase-1 (sFlt-1) Levels | At 20-24 weeks, 32-34 weeks, and 36 weeks gestation
  Serum levels of soluble fms-like tyrosine kinase-1 (sFlt-1) measured by immunoassay
Placental Growth Factor (PlGF) Levels | At 20-24 weeks, 32-34 weeks, and 36 weeks gestation
  Serum levels of placental growth factor (PlGF) measured by immunoassay
sFlt-1/PlGF Ratio | At 20-24 weeks, 32-34 weeks, and 36 weeks gestation
  Ratio of soluble fms-like tyrosine kinase-1 to placental growth factor (sFlt-1/PlGF ratio) measured by immunoassay
Interleukin-6 (IL-6) Levels | At 20-24 weeks, 32-34 weeks, and 36 weeks gestation
  Serum levels of interleukin-6 (IL-6) measured by immunoassay
Incidence of Early-Onset Preeclampsia | From enrollment until 34 weeks gestation
  Development of preeclampsia before 34 weeks gestation (early-onset preeclampsia)
Incidence of Gestational Hypertension | From 20 weeks gestation until delivery (up to 40 weeks)
  New-onset hypertension (blood pressure ≥140/90 mmHg on two occasions at least 4 hours apart) after 20 weeks gestation without proteinuria or evidence of end-organ dysfunction
Rate of Spontaneous Preterm Birth | From enrollment until delivery, assessed up to 40 weeks gestation
  Spontaneous preterm labor resulting in delivery before 34 weeks gestation and before 37 weeks gestation
Incidence of Small for Gestational Age | At delivery
  Birth weight below the 3rd, 5th, and 10th percentile for gestational age based on standardized fetal growth charts (small for gestational age)
Perinatal Death | From enrollment until 28 days after delivery
  Miscarriage, intrauterine fetal death, or neonatal death within 28 days after birth attributed to preeclampsia or fetal growth restriction
Neonatal Complications and Therapy | From delivery until hospital discharge (up to 3 months)
  Composite of neonatal adverse outcomes including sepsis, intraventricular hemorrhage grade III-IV, necrotizing enterocolitis, respiratory distress syndrome (RDS), need for surfactant therapy, mechanical ventilation, blood transfusion, and admission to neonatal intensive care unit (NICU) with duration of stay
Placental Abruption | From enrollment until delivery (up to 40 weeks gestation)
  Premature separation of the placenta from the uterine wall before delivery

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Daskalakis, PhD, Study Chair — First Department of Obstetrics and Gynecology, Alexandra Hospital
Locations (1):
- First Department of Obstetrics and Gynecology, Alexandra Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided
The decision on individual participant data sharing will be made in accordance with institutional policies and ethical requirements. The data sharing plan will be finalized prior to study completion and publication of results.

REFERENCES:
- [Background] McLaughlin K, Baczyk D, Potts A, Hladunewich M, Parker JD, Kingdom JC. Low Molecular Weight Heparin Improves Endothelial Function in Pregnant Women at High Risk of Preeclampsia. Hypertension. 2017 Jan;69(1):180-188. doi: 10.1161/HYPERTENSIONAHA.116.08298. Epub 2016 Nov 13. PMID 27840330
- [Background] Cruz-Lemini M, Vazquez JC, Ullmo J, Llurba E. Low-molecular-weight heparin for prevention of preeclampsia and other placenta-mediated complications: a systematic review and meta-analysis. Am J Obstet Gynecol. 2022 Feb;226(2S):S1126-S1144.e17. doi: 10.1016/j.ajog.2020.11.006. Epub 2021 Apr 20. PMID 34301348
- [Background] Wright D, Wright A, Nicolaides KH. The competing risk approach for prediction of preeclampsia. Am J Obstet Gynecol. 2020 Jul;223(1):12-23.e7. doi: 10.1016/j.ajog.2019.11.1247. Epub 2019 Nov 13. PMID 31733203
- [Background] Magee LA, Brown MA, Hall DR, Gupte S, Hennessy A, Karumanchi SA, Kenny LC, McCarthy F, Myers J, Poon LC, Rana S, Saito S, Staff AC, Tsigas E, von Dadelszen P. The 2021 International Society for the Study of Hypertension in Pregnancy classification, diagnosis & management recommendations for international practice. Pregnancy Hypertens. 2022 Mar;27:148-169. doi: 10.1016/j.preghy.2021.09.008. Epub 2021 Oct 9. PMID 35066406
- [Background] Rolnik DL, Wright D, Poon LC, O'Gorman N, Syngelaki A, de Paco Matallana C, Akolekar R, Cicero S, Janga D, Singh M, Molina FS, Persico N, Jani JC, Plasencia W, Papaioannou G, Tenenbaum-Gavish K, Meiri H, Gizurarson S, Maclagan K, Nicolaides KH. Aspirin versus Placebo in Pregnancies at High Risk for Preterm Preeclampsia. N Engl J Med. 2017 Aug 17;377(7):613-622. doi: 10.1056/NEJMoa1704559. Epub 2017 Jun 28. PMID 28657417
- [Background] Magee LA, Nicolaides KH, von Dadelszen P. Preeclampsia. N Engl J Med. 2022 May 12;386(19):1817-1832. doi: 10.1056/NEJMra2109523. No abstract available. PMID 35544388